CLINICAL TRIAL: NCT03806296
Title: Delayed Sleep Phase and Risk for Adolescent Substance Use
Brief Title: Delayed Sleep Timing in Teens Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brant Hasler, Assistant Professor of Psychiatry, Psychology, and Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19030063; R01DA044143 (NIH)
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Delayed Sleep Phase
Keywords: sleep; circadian; adolescence; substance use; reward; impulse control
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study combines Laboratory, Experimental, and Longitudinal protocols. The study includes 2 initial groups (Early/Middle Sleep Timing and Late Sleep Timing) that all complete the initial Laboratory (baseline) protocol. The Late Sleep participants are also randomized to complete one of two arms (Manipulation or Control) in the Experimental (intervention) protocol. The Early/Mid Sleep group does not complete the Experimental protocol. Finally, participants are also follow-up assessments through the life of the grant in the Longitudinal protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manipulation (Experimental): Participants who reported a weekend bedtime ≥ 1 AM.
  Completed both a 1-week baseline period (T1) and a 2-week experimental period (T2).
  During the 2-week experimental period, participants were asked to adhere to the following:
  * Sleep scheduling--advance bedtime by 1.5 hours ( + sleep duration)
  * Decrease evening blue light exposure via blue blocker goggles (2 h before bed)
  * Increase morning bright light exposure via bright light goggles (30 m after rise)
  * Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
  Interventions: Other: Increase morning bright light; Other: Decrease evening blue light; Behavioral: Sleep scheduling; Behavioral: Monitor sleep, mood, and substance use
- Control (Active Comparator): Participants who reported a weekend bedtime ≥ 1 AM.
  Completed both a 1-week baseline period (T1) and a 2-week experimental period (T2).
  During the 2-week experimental period, participants were asked to adhere to the following:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
  Interventions: Behavioral: Monitor sleep, mood, and substance use
- Early/Middle Sleep Timing (No Intervention): Participants who report a weekend bedtime <1AM. Participants completed only the 1-week baseline observational protocol (T1)

INTERVENTIONS:
Other: Increase morning bright light — Participants will wear Re-Timer bright glasses for 30 minutes each morning
  Arms: Manipulation
Other: Decrease evening blue light — Participants will wear tinted glasses that block blue wavelength light for 2 hours before bed
  Arms: Manipulation
Behavioral: Sleep scheduling — Participants will advance their weekday bedtime and maintain their weekday risetime on weekends
  Arms: Manipulation
Behavioral: Monitor sleep, mood, and substance use — Participants will monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraphy
  Arms: Control; Manipulation

SUMMARY:
This study will (1) comprehensively characterize the substance use disorder (SUD) risk profile associated with adolescent Delayed Sleep Phase (DSP), and (2) probe whether SUD risk is diminished by altering sleep/circadian timing.

DETAILED DESCRIPTION:
Mounting evidence indicates that delayed sleep phase (DSP) may confer risk for adolescent substance use (SU) and SUDs. However, the exact nature of this link and the mechanisms underlying it remain unclear. Circadian misalignment, a mismatch between late sleep hours and early school start times, is a compelling potential contributor to elevated SU in adolescent DSP with plausible neurobehavioral mechanisms. The investigators hypothesize that DSP-associated circadian misalignment decreases impulse control and increases reward sensitivity, thereby increasing SUD risk.

This study will, for the first time, (1) comprehensively characterize the SUD risk profile associated with adolescent DSP, and (2) probe whether SUD risk is diminished by altering sleep/circadian timing. The study will assess both established markers of SUD risk and putative neurobehavioral mechanisms (impulsivity and reward sensitivity). Specifically, the investigators will employ a comprehensive, multi-method approach to examining DSP's role in SUD risk, combining laboratory, experimental, and longitudinal studies. The investigators will recruit a sample of 150 eleventh and twelfth graders (16-19 y/o), divided between 100 DSP and 50 normal phase teens. The investigators will focus on cannabis and alcohol use given their prevalent use in adolescents and evident links to DSP.

In the laboratory study, the investigators will compare a group of DSP adolescents to a group of normal phase adolescents on behavioral and neuroimaging (fMRI) tasks tapping impulsivity and reward sensitivity, as well as a circadian phase assessment.

In the experimental study, the investigators will probe whether stabilizing circadian phase in the DSP group (n=100) by using sleep scheduling and chronotherapeutic approaches (i.e., dim light in the evening and bright light in the morning) improves sleep and neurobehavioral function relevant to SUD risk.

NOTE: When this ClinicalTrials.gov protocol was initially submitted, there were some mistakes made. The initial submission focused only on the Experimental study, which thus only included the "DSP group" (aka Late Sleep Timing group), and thus out the Laboratory study along with the "normal phase group" (aka Early/Middle Sleep Timing group). At that time, we also only listed a limited range of the primary outcomes listed in the funded grant, inadvertently leaving out several primary outcomes (weekday sleep duration - actigraph, circadian timing - dim light melatonin onset, neural correlates of reward receipt, and baseline cannabis and alcohol use). Finally, we mistakenly listed cannabis use from the Longitudinal protocol as a secondary outcome when it was actually an exploratory outcome in the funded grant, and thus we removed it.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-19 years
* Currently in 11th or 12th grade and enrolled in a traditional high-school; or cyber school with synchronous classes (not home-schooled)
* Physically and psychiatrically healthy, as determined by instruments described below
* Provision of written informed consent and assent

Additional inclusion criterion for Experimental protocol

* Meets operational definition of delayed sleep phase (DSP; weekend bedtime ≥1 AM)

Exclusion Criteria:

* Significant or unstable acute or chronic medical conditions
* Past or current bipolar disorder or psychotic disorder
* Past or current substance use disorder other than alcohol use disorder or cannabis use disorder
* Past month recreational drug use other than alcohol, cannabis, and nicotine
* Current syndromal sleep disorders other than insomnia and delayed sleep phase disorder
* Medications that interfere with sleep and/or reward function (antidepressants, and stimulants prescribed for ADHD are permitted)
* Conditions that would interfere with the MRI procedures (e.g., non-removal ferromagnetic devices)

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant P Hasler, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the surrounding community using flyers, postings on Pitt+Me (a registry for clinical and translational science research) and Read Green, word-of-mouth referrals, social media (Facebook/Instagram, Snapchat, YouTube, Spotify), Peach Jar (an online source for distributing flyers to schools), bus or church advertisements, local teen agencies, and school recruitment (contacting guidance counselors, teachers, and administrative employees).
Pre-assignment Details: The 142 enrolled participants include individuals who consented to the study, were randomized to a group, and completed a limited battery of baseline assessments during that consent/diagnostic interview visit, but did not necessarily continue on into the "Laboratory" (Baseline/T1) protocol.
Groups:
- Early/Middle Sleep Timing: Participants who reported a weekend bedtime <1AM.
  This group completed the T1 Baseline (aka Laboratory) phase and Longitudinal phase.
  Participants were asked to complete the following during a 7-day T1 Baseline phase:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the 7 days, participants were asked to complete an overnight visit in the sleep lab.
  After T1, participants entered the Longitudinal phase, during which they completed periodic self-report follow-ups through the life of the grant (every 2 months for the first 6 months, biannual after that up through 60 months).
- Late Sleep Timing - Control: Participants who reported a weekend bedtime ≥ 1 AM. This group completed the T1 Baseline (aka Laboratory) phase, T2 Post-Manipulation (aka Experimental) phase, and Longitudinal phase.
  Participants were asked to complete the following during a 7-day T1 Baseline phase:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph≥ At the conclusion of the 7 days, participants were asked to complete an overnight visit in the sleep lab.
  Next, the participants completed the 2-week T2 Post-Manipulation phase, during which they were asked to adhere to the following:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the ~2 weeks, participants were asked to complete an overnight visit in the sleep lab.
  After T2, participants entered the Longitudinal phase, during which they completed periodic self-report follow-ups through the life of the grant (every 2 months for the first 6 months, biannual after that up through 60 months).
- Late Sleep Timing - Manipulation: Participants who reported a weekend bedtime ≥ 1 AM. This group completed the T1 Baseline (aka Laboratory) phase, T2 Post-Manipulation (aka Experimental) phase, and Longitudinal phase.
  Participants were asked to complete the following during a 7-day T1 Baseline phase:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph≥ At the conclusion of the 7 days, participants were asked to complete an overnight visit in the sleep lab.
  Next, the participants completed the 2-week T2 Post-Manipulation phase, during which they were asked to adhere to the following:
  * Sleep scheduling--advance bedtime by 1.5 hours ( + sleep duration)
  * Decrease evening blue light exposure via blue blocker goggles (2 h before bed)
  * Increase morning bright light exposure via bright light goggles (30 m after rise)
  * Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the ~2 weeks, participants were asked to complete an overnight visit in the sleep lab.
  After T2, participants entered the Longitudinal phase, during which they completed periodic self-report follow-ups through the life of the grant (every 2 months for the first 6 months, biannual after that up through 60 months).
Period: T1: Laboratory: 1 Week
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Started (These include participants who consented to the study and completed a limited battery of baseline assessments during that consent/diagnostic interview visit, but did not necessarily continue on into the "Laboratory" (Baseline/T1) protocol.) | 56 | 42 | 44
Completed | 42 | 40 | 40
Not Completed | 14 | 2 | 4
Not completed — Withdrawal by Subject | 6 | 1 | 3
Not completed — Lost to Follow-up | 7 | 1 | 1
Not completed — Investigator withdrawn due to ineligibility learned post-enrollment. | 1 | 0 | 0
Period: T2: Experimental: 2 Weeks
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Started | 0 (The Early/Mid Sleep group did not complete the T2 Experimental protocol by design.) | 40 | 40
Completed | 0 | 38 | 38
Not Completed | 0 | 2 | 2
Period: Longitudinal Phase: 6 - 60 Months
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Started | 42 (Early/Middle Sleep participants did not complete T2 (by design), but the number of participants starting the Longitudinal protocol *does* match those continuing from T1.) | 40 (Although 2 participants of the 40 participants who started T2 did not finish all of the T2 protocol, they were all eligible to continue onto the Longitudinal protocol, which is why 40 participants started the Longitudinal protocol) | 38
Completed | 37 | 30 | 25
Not Completed | 5 | 10 | 13

BASELINE CHARACTERISTICS:
Population: The numbers in this section include all participants who consented, were determined eligible and interested, and started the Laboratory (baseline/T1) protocol (completed at least one day of the at-home actigraphy assessment).
Groups:
- Early/Middle Sleep Timing: Group definition: Participants who report a weekend bedtime <1AM.
  Also known as the Laboratory protocol.
  Participants are asked to complete the following during a 7-day baseline period:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the 7 days, participants are asked to complete an overnight visit in the sleep lab.
- Late Sleep Timing - Control; Late Sleep Timing - Manipulation: Group definition: Participants who reported a weekend bedtime ≥ 1 AM.
  Participants were randomized into either the Manipulation or Control Group.
  Also known as the Laboratory Protocol.
  Participants are asked to complete the following during a 7-day baseline period:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph≥ At the conclusion of the 7 days, participants are asked to complete an overnight visit in the sleep lab.
- Total: Total of all reporting groups
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation | Total
Number analyzed (Participants) | 42 | 40 | 40 | 122
Age, Continuous [Mean (Standard Deviation); unit: Age (in years)] | 17.4 (0.64) | 17.6 (0.55) | 17.4 (0.74) | 17.5 (0.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 26 | 76
  Male | 14 | 18 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 3 | 9
  Not Hispanic or Latino | 40 | 36 | 37 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 4 | 19
  White | 32 | 29 | 35 | 96
  More than one race | 1 | 3 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Weekday Sleep Duration - Actigraphy
Description: Total Sleep Time as determined by wrist actigraphy data (averaged across weekdays during 1 week of T1 and during 2 weeks of T2)
Time Frame: T1 (1 Week), T2 (2 Weeks)
Population: The numbers displayed in this section include the usable actigraph data collected for participants during T1. Early/Mid Sleep group only assessed at T1.
Measure: Mean (Standard Deviation); unit: Number of hours
Groups:
- Early/Middle Sleep Timing: Participants who report a weekend bedtime <1AM.
- Late Sleep Timing - Control: Group Definition: Participants who report a weekend bedtime >= 1AM and were randomized to the Control group for the Experimental protocol (T2)
  During the Experimental protocol, the Control group was asked to adhere to the following:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
- Late Sleep Timing - Manipulation: Group Definition: Participants who report a weekend bedtime >= 1AM and were randomized to the Manipulation group for the Experimental protocol (T2)
  During the Experimental protocol, the Manipulation group was asked to adhere to the following:
  * Sleep scheduling--advance bedtime by 1.5 hours ( + sleep duration)
  * Decrease evening blue light exposure via blue blocker goggles (2 h before bed)
  * Increase morning bright light exposure via bright light goggles (30 m after rise)
  * Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 42 | 40 | 39
Number of hours
  T1 | 6.309 (1.07) | 5.866 (0.963) | 5.880 (0.765)
  T2: number analyzed (Participants) | 0 | 38 | 38
  T2 |  | 5.845 (0.817) | 6.554 (0.801)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; For these Aim 1 analyses comparing the Early/Middle vs Late Sleep groups, the Late Sleep-Control and Late Sleep-Manipulation were combined into a single Late Sleep group. We used a linear regression model to test the effect of group (Early/Mid vs Late) on each a priori outcome, accounting for age and sex; Test type: Superiority; p = 0.018, Regression, Linear; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.77 to -0.07]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; For Aim 2, this mixed effect model tested the effect of group (Control vs Manipulation) on changes in each a priori outcome, accounting for group, timepoints, and sex; Test type: Superiority; p = 0.001, Mixed Models Analysis; Time X Group interaction = 0.67, 95% CI 2-sided [0.28 to 1.07]

2. Primary Outcome: Circadian Timing - Dim Light Melatonin Onset
Description: Circadian Timing as determined by dim light melatonin onset (DLMO) assessed during saliva sampling using the 4pg/ml threshold.
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday.
Population: The numbers displayed in this section include the usable data collected during the saliva sampling protocol at T1 overnight visits. Early/Mid Sleep group only assessed at T1.
Measure: Mean (Standard Deviation); unit: Clock Time (24-hour clock)
Groups:
- Early/Middle Sleep Timing: Group definition: Participants who report a weekend bedtime <1AM. Only complete the 1-week Laboratory protocol (T1)
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 38 | 36 | 40
Clock Time (24-hour clock)
  T1 | 20.707 (1.112) | 21.849 (1.395) | 21.789 (1.228)
  T2: number analyzed (Participants) | 0 | 31 | 34
  T2 |  | 22.038 (1.501) | 21.194 (1.355)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [0.61 to 1.59]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Time X Group interaction = -0.76, 95% CI 2-sided [-1.09 to -0.43]

3. Primary Outcome: Circadian Alignment
Description: Circadian alignment is operationalized as the interval between the dim light melatonin onset (DLMO) and sleep midpoint based on the prior two nights of actigraphy data.
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday. Based on DLMO assessed on weeknight lab overnight visit, and including the two nights of actigraphy data prior to the lab visit.
Population: The numbers displayed in this section include the participants with usable data collected during (1) the saliva sampling protocol at T1 overnight visits and (2) the actigraphy protocol in the two nights prior to the T1 visit. Early/Mid Sleep group only assessed at T1.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Early/Middle Sleep Timing: Group definition: Participants who report a weekend bedtime <1AM. Only completed the 1-week Observational protocol (T1)
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 38 | 36 | 39
Hours
  T1 | 6.071 (1.111) | 5.798 (1.142) | 5.937 (1.071)
  T2: number analyzed (Participants) | 0 | 36 | 39
  T2 |  | 5.910 (1.463) | 5.586 (1.243)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.365, Regression, Linear; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.64 to 0.24]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.067, Mixed Models Analysis; Time X Group interaction = -0.43, 95% CI 2-sided [-0.88 to 0.03]

4. Primary Outcome: Reward Motivation (Behavioral)
Description: Adjusted average pumps on Balloon Analogue Risk Task, a computerized measure of risk taking behavior in participants are presented with a series of balloons and offered the chance to earn money by pumping each balloon up by clicking a button. The adjusted average only includes non-burst trials.
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday.
Population: The numbers displayed in this section include the usable behavioral computer task data collected at T1 overnight visits. Early/Mid Sleep group only assessed at T1.
Measure: Mean (Standard Deviation); unit: Adjusted Average Number of pumps
Groups:
- Late Sleep Timing - Control: Group Definition: Participants who report a weekend bedtime >=1AM and were randomized to the Control group for the Experimental protocol (T2)
  During the Experimental protocol, the Control group was asked to adhere to the following:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 42 | 38 | 40
Adjusted Average Number of pumps
  T1 | 32.609 (13.274) | 37.696 (15.364) | 34.448 (14.416)
  T2: number analyzed (Participants) | 0 | 31 | 34
  T2 |  | 43.961 (13.508) | 34.117 (11.244)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.234, Regression, Linear; Mean Difference (Final Values) = 3.32, 95% CI 2-sided [-2.18 to 8.82]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; For Aim 2, this mixed effect model tested the effect of group (Control vs Manipulation) on changes in each a priori outcome, accounting for group, timepoint, and sex; Test type: Superiority; p = 0.018, Mixed Models Analysis; Time X Group interaction = -6.15, 95% CI 2-sided [-11.25 to -1.06]

5. Primary Outcome: Behavioral Inhibition
Description: Accuracy on Cued Go/No-Go Task, specifically correct response (withholding response) on No-Go trials following an incongruent Go cue
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Proportion accurate responses out of 1
Groups:
- Late Sleep Timing - Control: Group Definition: Participants who report a weekend bedtime < 1AM and were randomized to the Control group for the Experimental protocol (T2)
  During the Experimental protocol, the Control group was asked to adhere to the following:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 42 | 37 | 40
Proportion accurate responses out of 1
  T1 | 0.910 (0.108) | 0.891 (0.096) | 0.846 (0.124)
  T2: number analyzed (Participants) | 0 | 34 | 35
  T2 |  | 0.861 (0.131) | 0.829 (0.155)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.024, Regression, Linear; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [0.07 to 0.94]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.660, Mixed Models Analysis; Time X Group interaction = -0.10, 95% CI 2-sided [-0.55 to 0.35]

6. Primary Outcome: Neural Correlates of Reward Anticipation
Description: Activation within the reward network during the Monetary Incentive Delay task. Specifically, activation is defined as bold signal in regions of the reward network (from NeuroSynth) on reward anticipation trials (large reward) versus neutral (no money) trials. Higher values represent increased reactivity to reward, as compared to neutral trials.
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday.
Population: The numbers displayed in this section include the usable fMRI task data collected at the T1 visit. Early/Mid Sleep group only assessed at T1.
Measure: Mean (Standard Deviation); unit: percent signal change
Groups:
- Late Sleep Timing - Manipulation: During the Experimental protocol, the Manipulation group was asked to adhere to the following:
  * Sleep scheduling--advance bedtime by 1.5 hours ( + sleep duration)
  * Decrease evening blue light exposure via blue blocker goggles (2 h before bed)
  * Increase morning bright light exposure via bright light goggles (30 m after rise)
  * Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 37 | 32 | 34
percent signal change
  T1 | 0.040 (0.086) | 0.027 (0.123) | 0.074 (0.132)
  T2: number analyzed (Participants) | 0 | 29 | 31
  T2 |  | 0.007 (0.125) | 0.030 (0.087)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.592, Regression, Linear; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.03 to 0.06]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.550, Mixed Models Analysis; Time X Group interaction = -0.03, 95% CI 2-sided [-0.11 to 0.06]

7. Primary Outcome: Neural Correlates of Reward Receipt
Description: Monetary Incentive Delay Task: Win Outcome vs No Win contrast within the reward network (from Neurosynth). Higher values represent increased reactivity to reward wins, as compared to neutral trials.
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 37 | 33 | 35
percent signal change
  T1 | -0.009 (0.103) | -0.028 (0.135) | -0.019 (0.139)
  T2: number analyzed (Participants) | 0 | 28 | 32
  T2 |  | 0.009 (0.100) | -0.008 (0.074)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.550, Regression, Linear; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.07 to 0.04]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.556, Mixed Models Analysis; Time X Group interaction = -0.02, 95% CI 2-sided [-0.10 to 0.06]

8. Primary Outcome: Neural Correlates of Impulse Control
Description: Activation within the Executive Control Network during the Stop Signal Task. Specifically, activation is defined as bold signal in regions of the Executive Control Network on unsuccessful Stop trials versus successful Go trials. Higher values represent increased activity to unsuccessful Stop versus successful Go trials.
Time Frame: Overnight visits at end of T1 (1 Week) and T2 (2 Weeks). Always occurred on a Wednesday or Thursday.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 26 | 27 | 35
percent signal change
  T1 | 0.047 (0.080) | 0.066 (0.063) | 0.070 (0.072)
  T2: number analyzed (Participants) | 0 | 24 | 19
  T2 |  | 0.049 (0.071) | 0.054 (0.078)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.124, Regression, Linear; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.06]
Statistical Analysis 2: Comparison: Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.925, Mixed Models Analysis; Time X Group interaction = 0.00, 95% CI 2-sided [-0.05 to 0.06]

9. Primary Outcome: Cannabis Use
Description: Days of cannabis use based on timeline followback interview administered during baseline interview during consent/diagnostic interview visit.
Time Frame: Days of cannabis use in 3 months prior to baseline.
Population: The numbers in this section include all participants who consented, were determined eligible and interested, and started the Laboratory (T1) protocol.
Measure: Mean (Standard Deviation); unit: Days of use
Groups:
- Late Sleep Timing - Control: Group Definition: Participants who report a weekend bedtime >= 1AM and were randomized to the Control group for the Experimental protocol (T2)
- Late Sleep Timing - Manipulation: Group Definition: Participants who report a weekend bedtime >= 1AM and were randomized to the Manipulation group for the Experimental protocol (T2)
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 42 | 40 | 40
Days of use | 2.167 (5.708) | 3.200 (10.115) | 2.148 (6.928)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; For these Aim 1 analyses comparing the Early/Middle vs Late Sleep groups, the Late Sleep-Control and Late Sleep-Manipulation were combined into a single Late Sleep group. We used a Poisson generalized linear model (GLM) to test the effect of group (Early/Mid vs Late) on a binary cannabis use outcome (yes/no in the past 3 months), accounting for age and sex; Test type: Superiority; p = 0.42, Poisson GLM with robust standard error; Risk Ratio (RR) = 0.752, 95% CI 2-sided [0.374 to 1.513] — Early/Middle Sleep group was the reference group (lower RR indicates less likelihood of cannabis use in the Late Sleep group)

10. Primary Outcome: Alcohol Use
Description: Days of alcohol use based on timeline followback interview administered during baseline interview during consent/diagnostic interview visit.
Time Frame: 3 months prior to baseline, based on timeline followback interview.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Days of use
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
Number analyzed (Participants) | 42 | 40 | 40
Days of use | 0.381 (0.697) | 1.275 (2.961) | 1.325 (2.515)
Statistical Analysis 1: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; For these Aim 1 analyses comparing the Early/Middle vs Late Sleep groups, the Late Sleep-Control and Late Sleep-Manipulation were combined into a single Late Sleep group. We used a Poisson generalized linear model (GLM) to test the effect of group (Early/Mid vs Late) on a binary alcohol use outcome (yes/no in the past 3 months), accounting for age and sex; Test type: Superiority; p = 0.461, Poisson GLM with robust standard error; Risk Ratio (RR) = 1.236, 95% CI 2-sided [0.704 to 2.171] — Early/Middle Sleep group was the reference group (higher RR indicates higher likelihood of alcohol use in the Late Sleep group)
Statistical Analysis 2: Comparison: Early/Middle Sleep Timing vs Late Sleep Timing - Control vs Late Sleep Timing - Manipulation; For these Aim 1 analyses comparing the Early/Middle vs Late Sleep groups, the Late Sleep-Control and Late Sleep-Manipulation were combined into a single Late Sleep group. We used a negative binomial GLM to test the effect of group (Early/Mid vs Late) on days of alcohol use, accounting for age and sex; Test type: Superiority; p = 0.007, negative binomial glm; Incident Rate Ratio = 3.29, 95% CI 2-sided [1.36 to 7.90] — Early/Middle Sleep group was the reference group (higher IRR indicates greater days of alcohol use in the Late Sleep group than in the Early/Middle Sleep group)

ADVERSE EVENTS:
Time Frame: 1 - 3 weeks (1 week for Early/Mid Sleep participants; 3 weeks for Late Sleep participants)
Description: Adverse events were monitored during the T1/Baseline/Laboratory and T2/Post-Manipulation/Experimental phases, and not during the Longitudinal phase.
Groups:
- Early/Middle Sleep Timing: Participants who report a weekend bedtime <1AM.
  Participants are asked to complete the following during a 7-day baseline period:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the 7 days, participants are asked to complete an overnight visit in the sleep lab.
- Late Sleep Timing - Control: Participants who reported a weekend bedtime ≥ 1 AM.
  Participants are asked to complete the following during a 7-day baseline period:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph≥ At the conclusion of the 7 days, participants are asked to complete an overnight visit in the sleep lab.
  For the next ~2 weeks, participants will asked to adhere to the following:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the ~2 weeks, participants are asked to complete an overnight visit in the sleep lab.
- Late Sleep Timing - Manipulation: Participants who reported a weekend bedtime ≥ 1 AM.
  Participants are asked to complete the following during a 7-day baseline period:
  - Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph≥ At the conclusion of the 7 days, participants are asked to complete an overnight visit in the sleep lab.
  For ~2 weeks, participants will be asked to adhere to the following:
  * Sleep scheduling--advance bedtime by 1.5 hours ( + sleep duration)
  * Decrease evening blue light exposure via blue blocker goggles (2 h before bed)
  * Increase morning bright light exposure via bright light goggles (30 m after rise)
  * Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph At the conclusion of the ~2 weeks, participants are asked to complete an overnight visit in the sleep lab.
Arm/Group | Early/Middle Sleep Timing | Late Sleep Timing - Control | Late Sleep Timing - Manipulation
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT03806296/Prot_SAP_000.pdf